CLINICAL TRIAL: NCT00581802
Title: Cohort Study to Understand Resistance and HIV Eradication (CURE): Observational Studies of Antiretroviral Drug Treatment Success and Failure
Brief Title: HIV Resistance and Treatment Strategies
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Vanderbilt University School of Medicine (Other)
Responsible Party: Principal Investigator, Richard T D'Aquila, Professor of Medicine, Vanderbilt University, National Institute of Allergy and Infectious Diseases (NIAID)
Other Study IDs: 1R43AI062473-01 (NIH); CURE
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: CD4-Positive T-Lymphocytes; Treatment Naive; Latent HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, white cells, and whole blood

GROUPS / COHORTS (5):
- 1: Intensively studied participants initiating potentially suppressive drug therapy. Group 1 participants may undergo optional leukapheresis. Group 1 participants may decline to be in the leukapheresis group at any time and will be given the option of continuing in the blood draw group or withdrawing from the study. If specimens are not obtained for any reason at any visit, Group 1 participants will default to either Group 3 or Group 4.
- 2: Intensively studied, well-suppressed participants on HAART. Participants in Group 2 may undergo optional leukapheresis. Group 2 participants may decline to be in the leukapheresis group at any time and will be given the option of continuing in the blood draw group or withdrawing from the study. If specimens are not obtained for any reason at any visit, Group 2 participants will default to either Group 3 or Group 4.
- 3: Nonintensively studied participants initiating potentially suppressive drug therapy
- 4: Nonintensively studied well-suppressed participants on HAART
- 5: Intensively studied participants who are currently participating in the Merck Expanded Access Program and receiving raltegravir. Participants in Group 5 may undergo optional leukapheresis. Group 5 participants may decline to be in the leukapheresis group at any time and will be given the option of continuing in the blood draw group or withdrawing from the study. If specimens are not obtained for any reason at any visit, Group 5 participants will default to either Group 3 or Group 4.

SUMMARY:
The purpose of this observational study is to characterize which immune system cells hide the latent reservoir of HIV by counting the number of latent HIV in different subsets of CD4 cells. Observations will also be made on other possible mechanisms of HIV persistence by looking at cellular factors such as APOBEC3 and drug transporters. The purpose of this study is to develop new strategies to reduce and possibly eliminate the latent reservoir in HIV infected adults.

DETAILED DESCRIPTION:
Memory CD4 cells may provide a reservoir of latent HIV that cannot be completely eliminated using currently available anti-HIV medications. The overall goal of this observational study is to develop new strategies to eliminate the latent HIV reservoir in HIV infected individuals. CD4-cell subsets, cellular anti-HIV factors, and cellular drug transporters will be observed to determine which resting memory cells hide latent HIV and to determine the mechanisms responsible for the persistence of the latent HIV reservoir.

This study will last for at least 3 years. The screening visit will include medical history, contact information, urine collection, and a physical exam. Participants will be assigned to one of five groups:

* Group 1 will consist of intensively studied adults initiating potentially suppressive drug therapy. At the screening visit, Group 1 participants will be given the option to either undergo blood draws or leukapheresis for all visits.
* Group 2 will consist of intensively studied, well-suppressed adults on highly active antiretroviral therapy (HAART). At the screening visit, Group 2 participants will be given the option to either undergo blood draws or leukapheresis for all visits.
* Group 3 will consist of nonintensively studied adults initiating potentially suppressive drug therapy. Group 3 participants will undergo blood draws at all visits.
* Group 4 will consist of nonintensively studied, well-suppressed adults on HAART. Group 4 participants will undergo blood draws at all visits.
* Group 5 will consist of participants who are currently in the Merck Expanded Access Program receiving raltegravir. At the screening visit, Group 5 participants will be given the option to either undergo blood draws or leukapheresis for all visits.

For all participants undergoing blood draws only, visits will occur every 3 months for about 3 years. For patients undergoing leukapheresis, visits will occur every 6 months for about 3 years. At each visit, blood collection, documentation of current HAART, and updating of contact information will occur. Participants are encouraged to provide additional blood samples to be stored at all visits.

Participants in Groups 1, 2, or 5 may decline to be in the leukapheresis group at any time and will be given the option of continuing in the blood draw group or withdrawing completely from the study. If specimens are not obtained for any reason at any visit, participants in Groups 1, 2, or 5 will default to either Group 3 or Group 4. Antiretroviral medications will not be provided by this study.

ELIGIBILITY:
Inclusion Criteria for Groups 1 and 3:

* HIV infected
* Antiretroviral therapy (ART) naive OR a history of treatment with highly active antiretroviral therapy (HAART), a currently detectable viral load greater than 500 copies/ml, about to begin second or later potentially suppressive antiretroviral regimen, and must meet the following two requirements:

  1. Viral load less than 50 copies/ml on the immediately prior regimen with less than 50 copies/ml measured on at least two visits during prior ART
  2. Viral load greater than 500 copies/ml on two consecutive visits and a history of failure during prior lamivudine- or emtricitabine-containing ART

Exclusion Criteria for Groups 1 and 3:

* History of treatment with any two of the following: darunavir, tipranavir, or enfuvirtide
* Self-reported or clinician-reported nonadherence to earlier ART
* Current substance abuse that, in the opinion of the investigator, will increase the risk of nonadherence
* Weight less than 110 lbs
* Blood transfusion within the 6 months prior to study entry
* Platelets less than 50 cells/mm3
* International normalized ratio (INR) greater than 2.0 if participants are on warfarin
* Heart disease with recent angina or myocardial infarction (MI) within 1 year prior to study entry
* Hematocrit 28% or less OR hemoglobin 8.0 g/dl or less
* Prior ART that included only one or two drugs
* Pregnancy

Inclusion Criteria for Groups 2 and 4:

* HIV infected
* Currently on HAART with an undetectable viral load of less than 50 copies/ml for 12 months prior to study entry (at least two measures). If the participant is on the second or later regimen of HAART, the previous regimen must have contained lamivudine or emtricitabine.

Exclusion Criteria:

* Viral load "blip" greater than 2,000 copies/ml during current suppressive regimen
* Consistent low level viral load (between 50 and 2,000 copies/ml) during current regimen
* Change in currently suppressing HAART before study entry
* Self-reported or clinician-reported nonadherence to earlier antiretroviral regimens
* Current substance abuse that, in the opinion of the investigator, will increase the risk of nonadherence
* Weight less than 110 lbs
* Blood transfusion within the 6 months prior to study entry
* Platelets less than 50 cells/mm3
* INR greater than 2.0 if participants are on warfarin
* Heart disease with recent angina or MI within 1 year prior to study entry
* Hematocrit 28% or less OR hemoglobin 8.0 g/dl or less
* Prior ART that included only one or two drugs
* Pregnancy

Inclusion Criteria for Group 5:

* HIV infected
* Currently taking or about to begin raltegravir with optimized background HAART

Exclusion Criteria:

* Current substance abuse that, in the opinion of the investigator, will increase the risk of nonadherence
* Weight less than 110 lbs
* Blood transfusion 6 months prior to study entry
* Platelets less than 50/mm3
* INR greater than 2.0 if participants are on warfarin
* Heart disease with recent angina or MI within 1 year prior to study entry
* • Hematocrit 28% or less OR hemoglobin 8.0 g/dl or less
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Comprehensive Care Clinic, a clinic that provides care exclusively to HIV patients from middle Tennessee and surrounding states. Participants are screened and identified with the inclusion and exclusion criteria from the computerized medical records system. If the medical charts are tagged, the study nurse will speak to the selected participant at the participant's following appointment.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-01; Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Establishment of a longitudinal, observational cohort of chemotherapeutically suppressed HIV participants to study cellular and virologic characteristics that enable HIV latency | At the end of the study

SECONDARY OUTCOMES:
Characterization of memory CD4 cell subsets isolated from chemotherapeutically suppressed participants | At the end of the study
Quantification of the amount of latent HIV in each memory cell type in chemotherapeutically suppressed participants | At the end of the study
Evidence of HIV evolution | At the end of the study
Characterization of certain proteins in memory CD4-cell subsets in chemotherapeutically suppressed participants | At the end of the study
Determination of the association of protein regulation with cellular toxicity and the latent HIV reservoir in chemotherapeutically suppressed participants | At the end of the study
Characterization of the effects of immune activation on the latent reservoir of HIV | At the end of the study
Determination of the role of drug transporters in chemotherapeutically suppressed patients | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. D'Aquila, MD, Principal Investigator — Vanderbilt University; Carey K. Hwang, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Comprehensive Care Clinic/Center for AIDS Research, Nashville, Tennessee, United States

REFERENCES:
- [Background] Noe A, Plum J, Verhofstede C. The latent HIV-1 reservoir in patients undergoing HAART: an archive of pre-HAART drug resistance. J Antimicrob Chemother. 2005 Apr;55(4):410-2. doi: 10.1093/jac/dki038. Epub 2005 Feb 22. PMID 15728140
- [Background] Pomerantz RJ. Reservoirs, sanctuaries, and residual disease: the hiding spots of HIV-1. HIV Clin Trials. 2003 Mar-Apr;4(2):137-43. doi: 10.1310/80jh-148k-nadq-u927. PMID 12671782
- [Background] Sedaghat AR, Siliciano JD, Brennan TP, Wilke CO, Siliciano RF. Limits on replenishment of the resting CD4+ T cell reservoir for HIV in patients on HAART. PLoS Pathog. 2007 Aug 31;3(8):e122. doi: 10.1371/journal.ppat.0030122. PMID 17784786
- [Background] Siliciano JD, Siliciano RF. A long-term latent reservoir for HIV-1: discovery and clinical implications. J Antimicrob Chemother. 2004 Jul;54(1):6-9. doi: 10.1093/jac/dkh292. Epub 2004 May 26. PMID 15163657